CLINICAL TRIAL: NCT01314898
Title: A Phase 1, Double-Blind (Sponsor-Open), Placebo- And Active-Controlled, Single Dose, Crossover Study To Assess Antimineralocorticoid Activity Of Oral Pf-03882845 In Healthy Subjects.
Brief Title: A Single Dose Study Of Antimineralocorticoid Activity Of PF-03882845 In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: B0171007; B0171007
Record Dates: First submitted 2011-03-03; First posted 2011-03-15 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2011-07

CONDITIONS: Healthy Volunteers
Keywords: Single dose; cross-over; active-control; placebo control; antimineralocorticoid activity
MeSH Terms: interventions — (3S,3aR)-2-(3-chloro-4-cyanophenyl)-3-cyclopentyl-3,3a,4,5-tetrahydro-2H-benzo(g)indazole-7-carboxylic acid; Spironolactone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental)
  Interventions: Drug: 3 mg PF-03882845; Drug: 10 mg PF-03882845; Drug: 30 mg PF-03882845; Drug: 100 mg PF-03882845; Drug: Spironolactone

INTERVENTIONS:
Drug: 3 mg PF-03882845 — 3 mg PF-03882845, single oral dose
Drug: 10 mg PF-03882845 — 10 mg PF-03882845, single oral dose
Drug: 30 mg PF-03882845 — 30 mg PF-03882845, single oral dose
Drug: 100 mg PF-03882845 — 100 mg PF-03882845, single oral dose
Drug: Spironolactone — 100 mg spironolactone, single oral dose

SUMMARY:
24-hr urinary sodium/potassium ratio will be a sensitive biomarker of antimineralocorticoid activity. The dose-response relationship of the antimineralocorticoid activity of PF-03882845 can be established following single oral doses.

ELIGIBILITY:
Inclusion Criteria:

* Male and/or female healthy volunteers, age 18 to 55 years. Females must be of non-childbearing potential.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).
* Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, diet restrictions and other trial procedures.

Exclusion Criteria:

* Subjects with a supine BP >140 mm Hg systolic or >90 mm Hg diastolic or <100 mm Hg systolic or <60 mm Hg diastolic based on the average of the triplicate
* Serum potassium >=5.1 mmol/L or <3.5 mmol/L at screening, confirmed by a single repeat if deemed necessary.
* Estimated GFR <60 mL/min/1.73 m2 using the Cockcroft-Gault formula measurement of the individual parameters following at least 5 minutes of rest at Screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2011-03; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Twenty-four hour urinary Na/K ratio (AUC(0-24)). | 0-24hr postdose per period

SECONDARY OUTCOMES:
Area Under the Curve(AUClast) from the time of dosing to the last data point of PF-03882845. | 0-24 hr post dose per period
Time of Maximum concentration(Tmax) of PF-03882845. | 0-24 hr post dose per period
Maximum concentration (Cmax) of PF-03882845. | 0-24 hr post dose per period
Safety and tolerability: Physical examinations, adverse event monitoring, clinical safety laboratory assessments, vital sign measurements and 12-lead ECGs. | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0171007&StudyName=A%20Single%20Dose%20Study%20Of%20Antimineralocorticoid%20Activity%20Of%20PF-03882845%20In%20Healthy%20Volunteers